CLINICAL TRIAL: NCT02903121
Title: Treatment of Unfavorable Bleeding Patterns in Contraceptive Implant Users
Acronym: Tamoxifen/BTB
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oregon Health and Science University (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Principal Investigator, Alison Edelman, Professor, OB/GYN, Oregon Health and Science University
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: OHSU IRB 16519
Record Dates: First submitted 2016-09-13; First posted 2016-09-16 (Estimated); Results first posted 2020-07-07 (Actual); Last update posted 2020-07-15 (Actual); Status verified 2020-07

CONDITIONS: Bleeding; Implants; Breakthrough Bleeding
Keywords: Unscheduled bleeding; Long acting contraception
MeSH Terms: conditions — Hemorrhage; Metrorrhagia | interventions — Tamoxifen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Tamoxifen (Experimental): Tamoxifen 10 mg (oral) twice daily for 7 days to be started following 3 consecutive days of bleeding
  Interventions: Drug: Tamoxifen; Drug: Tamoxifen (open label)
- Placebo (Placebo Comparator): Placebo (oral) twice daily for 7 days to be started following 3 consecutive days of bleeding
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tamoxifen — Tamoxifen 10 mg orally twice daily for 7 days. Treatment to be started after 3 consecutive days of bleeding and can be repeated every 30 days two more times in the first 90 days of the study
  Other Names: Nolvadex; Genox; Tamifen
  Arms: Tamoxifen
Drug: Placebo — Placebo orally twice daily for 7 days. Treatment to be started after 3 consecutive days of bleeding and can be repeated every 30 days two more times in the first 90 days of the study
  Arms: Placebo
Drug: Tamoxifen (open label) — Tamoxifen 10 mg orally twice daily for 7 days. Treatment to be started after 3 consecutive days of bleeding and can be repeated every 30 days two more times in the second 90 days of the study
  Other Names: Nolvadex; Genox; Tamifen
  Arms: Tamoxifen

SUMMARY:
The etonogestrel (ENG) subdermal contraceptive implant (ENG implant) is a highly effective method of preventing pregnancy, but it has bleeding side effects that make it unappealing for many women. The only study to demonstrate a sustained reduction in bleeding lasting for two months was the selective estrogen receptor modulator (SERM) tamoxifen in users of the levonogestrel (LNG) contraceptive implant. Based on the investigators encouraging preliminary data of tamoxifen and ENG implant users, the investigators plan to perform additional studies on the impact of tamoxifen on the breakthrough bleeding experience by ENG implant users.

DETAILED DESCRIPTION:
The investigators will perform a 2 phase trial for treatment of women experiencing frequent or prolonged bleeding while using the ENG contraceptive implant. The first phase will consist of a randomized, controlled, double blind placebo-controlled clinical trial over a 90-day reference period and the second phase will allow both study arms to receive open-label treatment over an additional 90-day reference period. The primary outcome of the study will be the total number of consecutive bleeding-free days in first 30 days from Day 1 of first treatment (TX1).

ELIGIBILITY:
Inclusion Criteria:

* English or Spanish speaking
* women aged 15-45 years of age
* Currently using the ENG-implant for at least 1 month and use proven on exam (palpation of implant at screening visit)
* Willing to continue using the implant for at least 6 months
* >7 days of continuous bleeding/spotting, or 2 or more episodes of bleeding/spotting in the last 30 days.
* Cellphone that is able to receive and respond to a daily text or email message .

Exclusion Criteria:

* Postpartum within six months
* post-abortion within six weeks
* currently pregnant
* currently breast-feeding
* undiagnosed abnormal uterine bleeding pre-dating placement of contraceptive implant
* bleeding dyscrasia
* anticoagulation use
* active cervicitis
* allergy to tamoxifen
* history of venous thromboembolism
* current or past breast or uterine malignancy
* use of medication contraindicated with tamoxifen (coumadin, letrozole, bromocriptine, rifampicin, aminoglutethimide, phenobarbital).

Ages: 15 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 109 (Actual)
Dates: Start 2017-01-20 (Actual); Primary Completion 2019-06-05 (Actual); Study Completion 2019-06-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- OHSU, Portland, Oregon, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Edelman AB, Kaneshiro B, Simmons KB, Hauschildt JL, Bond K, Boniface ER, Jensen JT. Treatment of Unfavorable Bleeding Patterns in Contraceptive Implant Users: A Randomized Controlled Trial. Obstet Gynecol. 2020 Aug;136(2):323-332. doi: 10.1097/AOG.0000000000003896. PMID 32649493

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Tamoxifen | Placebo
Started | 57 | 52
Completed | 34 | 38
Not Completed | 23 | 14

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Tamoxifen | Placebo | Total
Number analyzed (Participants) | 55 | 52 | 107
Age, Continuous [Mean (Standard Deviation); unit: Years] | 24.5 (5.1) | 23.4 (4.5) | 23.9 (4.8)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 55 | 52 | 107
  Male | 0 | 0 | 0
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 30 | 32 | 62
  Hispanic | 8 | 10 | 18
  Asian | 7 | 4 | 11
  Black | 1 | 2 | 3
  More than one | 7 | 4 | 11
  Other or unspecified | 2 | 0 | 2
Marital Status [Count of Participants; unit: Participants]
  Single or divorced | 13 | 18 | 31
  Partnered or Married | 42 | 34 | 76
Education [Count of Participants; unit: Participants]
  High school or less | 10 | 7 | 17
  College (any or more) | 45 | 45 | 90
Days of implant use at study entry [Mean (Standard Deviation); unit: Days] | 370.8 (267.7) | 469.1 (274.5) | 418.6 (274.2)

OUTCOME MEASURES:

1. Primary Outcome: Total Number of Consecutive Bleeding-free Days in First 30 Days From Day 1 of First Treatment (TX1)
Description: Bleeding free days in the first 30 days
Time Frame: Day 1 to Day 30
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 55 | 52
days | 18.5 (17) | 8.7 (8.4)

2. Secondary Outcome: Total Number of Bleeding Free Days Over the First 90 Day Reference Period From Day 1 of Treatment 1.
Description: bleeding free days in the first 90 days
Time Frame: Day 1 to Day 90
Measure: Median (Full Range); unit: days
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 46 | 42
days | 60 [18 to 84] | 52 [11 to 67]

3. Other Pre Specified Outcome: Total Number of Bleeding Free Days Over the Second 90 Day Reference Period From Day 1 of Treatment Number 4 to Day 90
Description: bleeding free days in the second 90 days
Time Frame: Day 1 of treatment number 4 to Day 90 (second 90 day reference period)
Measure: Median (Full Range); unit: days
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 39 | 42
days | 56 [6 to 81] | 67.5 [7 to 83]

4. Other Pre Specified Outcome: Patient Satisfaction With Bleeding Pattern
Description: Patient satisfaction with bleeding pattern. Assessed by visual analog scale to determine satisfaction with bleeding patterns on a scale of 0-100 mm, where 0 mm represents not satisfied at all and 100 mm is totally satisfied.
Time Frame: Day 1 of treatment 1 to day 180
Measure: Median (Full Range); unit: mm
Arm/Group | Tamoxifen | Placebo
Number analyzed (Participants) | 38 | 40
mm | 67.5 [0 to 100] | 54.25 [0.5 to 98]

ADVERSE EVENTS:
Time Frame: 180 day duration of study participation
Arm/Group | Tamoxifen | Placebo
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/52
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/52
Other Adverse Events (participants affected / at risk) | 45/55 | 12/52
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Tamoxifen (N=55) | Placebo (N=52)
Cramping, changes in menstrual fluid (Reproductive system and breast disorders) | 3 | 0
Fluid retention (Blood and lymphatic system disorders) | 10 | 1
Headache, migraine (Nervous system disorders) | 16 | 1
Hot flashes (Nervous system disorders) | 6 | 3
Mood changes (Psychiatric disorders) | 11 | 2
Nausea, Vomiting (Gastrointestinal disorders) | 5 | 2
Weakness, fatigue, dizziness (Nervous system disorders) | 6 | 1
Yeast infection, bacterial vaginosis (Reproductive system and breast disorders) | 5 | 0
Acne (Skin and subcutaneous tissue disorders) | 0 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2019-08-07): https://cdn.clinicaltrials.gov/large-docs/21/NCT02903121/Prot_001.pdf